CLINICAL TRIAL: NCT01189227
Title: A Phase III Study Evaluating the Role of Perioperative Chemotherapy in Patients With Potentially Resectable Hepatic Colorectal Metastases
Brief Title: Combination Chemotherapy Before or After Surgery in Treating Patients With Colorectal Cancer With Liver Metastases That Could Be Removed By Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to low accrual.
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP C-11; NSABP-C-11
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; adenocarcinoma of the colon; stage IV rectal cancer; adenocarcinoma of the rectum; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Postoperative chemotherapy (Experimental): Patients undergo hepatic resection. Beginning 31-56 days after surgery, patients receive mFOLFOX6 or FOLFIRI chemotherapy IV on day 1 over 3 hours. Patients receive an additional dose of fluorouracil over 46 hours using a portable pump. Treatment repeats every 2 weeks for 12 cycles.
  Interventions: Procedure: Postoperative chemotherapy
- Arm 2: Perioperative chemotherapy (Experimental): Patients receive mFOLFOX6 or FOLFIRI chemotherapy IV over 3 hours on day 1. Patients receive an additional dose of fluorouracil over 46 hours using a portable pump. Treatment repeats for every 2 weeks for 6 cycles. Patients then undergo hepatic resection. Beginning 31-56 days after surgery, patients receive an additional 6 cycles of mFOLFOX6 or FOLFIRI chemotherapy.
  Interventions: Procedure: Perioperative chemotherapy

INTERVENTIONS:
Procedure: Postoperative chemotherapy — Patients undergo hepatic resection. Beginning 31-56 days after surgery, patients receive mFOLFOX6 or FOLFIRI chemotherapy IV on day 1 over 3 hours. Patients receive an additional dose of fluorouracil over 46 hours using a portable pump. Treatment repeats every 2 weeks for 12 cycles.
  Arms: Arm 1: Postoperative chemotherapy
Procedure: Perioperative chemotherapy — Patients receive mFOLFOX6 or FOLFIRI chemotherapy IV over 3 hours on day 1. Patients receive an additional dose of fluorouracil over 46 hours using a portable pump. Treatment repeats for every 2 weeks for 6 cycles. Patients then undergo hepatic resection. Beginning 31-56 days after surgery, patients receive an additional 6 cycles of mFOLFOX6 or FOLFIRI chemotherapy.
  Arms: Arm 2: Perioperative chemotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to kill tumor cells or stop them from growing. Giving combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving combination chemotherapy after surgery may kill any remaining tumor cells. It is not yet known whether giving combination chemotherapy before and after surgery is more effective than giving combination chemotherapy after surgery.

PURPOSE: This randomized phase III trial is studying giving combination chemotherapy before and after surgery to see how well it works compared to giving combination chemotherapy after surgery in treating patients with colorectal cancer with liver metastases that could be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the difference in recurrence-free survival (RFS) of patients with potentially resectable hepatic colorectal metastases receiving perioperative (preoperative plus postoperative) adjuvant chemotherapy vs only postoperative adjuvant chemotherapy following liver resection for colorectal metastases.

Secondary

* To compare the proportion of patients between study arms who are R0 or R1 resected, alive, and free of recurrence at 6 months.
* To compare RFS between study arms in the cohort of patients event-free at 6 months.
* To compare overall survival between study arms.
* To evaluate the difference in R0 and combined R0 + R1 resection rates in patients receiving neoadjuvant therapy and those undergoing initial surgical resection.
* To compare the postoperative morbidity profile between study arms.
* To evaluate the safety and toxicity profile of postoperative and perioperative administration of chemotherapy and bevacizumab.

Tertiary

* To evaluate the relationship of baseline circulating tumor cells (CTC) to RFS.
* To evaluate the relationship of baseline CTC to R0 resection.
* To evaluate the relationship of pre-resection CTC in the preoperative therapy group only with RFS and R0 resection.

OUTLINE: This is a multicenter study. Patients are stratified by number of liver metastases (1-3 vs 4+), chemotherapy regimen* (mFOLFOX6 vs FOLFIRI), and synchronous** primary colorectal cancer (yes vs no). Patients are randomized to 1 of 2 treatment arms.

NOTE: *Patients who have not received previous oxaliplatin receive mFOLFOX6 chemotherapy comprising oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 46 hours on day 1. Patients who have received previous oxaliplatin receive FOLFIRI chemotherapy comprising irinotecan hydrochloride IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 46 hours on day 1.

NOTE: **Synchronous is defined as the detection (by imaging) of suspicious liver metastases within 90 days before or after the date of histologic diagnosis of the primary colon or rectal cancer.

* Arm 1 (postoperative): Patients undergo hepatic resection. Beginning 31-56 days after surgery, patients receive mFOLFOX6 or FOLFIRI chemotherapy IV on day 1 over 3 hours. Patients receive an additional dose of fluorouracil over 46 hours using a portable pump. Treatment repeats every 2 weeks for 12 courses.
* Arm 2 (perioperative): Patients receive mFOLFOX6 or FOLFIRI chemotherapy IV over 3 hours on day 1. Patients receive an additional dose of fluorouracil over 46 hours using a portable pump. Treatment repeats for every 2 weeks for 6 courses. Patients then undergo hepatic resection. Beginning 31-56 days after surgery, patients receive an additional 6 courses of mFOLFOX6 or FOLFIRI chemotherapy.

Blood and tumor tissue samples may be collected periodically for correlative studies.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal adenocarcinoma

  * Hepatic metastasis (no histologic confirmation required) and no evidence of extrahepatic metastatic disease within the past 4 weeks by one of the following imaging studies*:

    * PET/CT scan with contrast
    * PET scan AND CT scan with contrast
    * PET scan AND MRI with contrast
    * PET/CT scan without contrast AND MRI with contrast NOTE: *If findings noted in imaging study reports are equivocal, the determination of whether or not the findings represent extrahepatic disease will be at the investigator's discretion.
  * No history of or concurrent evidence of extrahepatic metastases

    * Patients with regional nodes that are suspicious on imaging and are associated with the primary colorectal tumor are eligible provided the nodes will be resected with the primary tumor after randomization
  * No radiographic evidence of metastases to portal lymph nodes (node > 1 cm in diameter) unless the node(s) are proven by biopsy to be negative
* No anal, small bowel, or appendiceal carcinoma
* No sarcoma, lymphoma, or carcinoid colorectal malignant diseases
* Within 4 weeks before randomization, the liver metastases must be determined by a hepatic surgeon to be resectable based on meeting both of the following criteria:

  * A complete resection can be performed in a single operation
  * There are ≥ 2 uninvolved contiguous segments of the liver
* Meets one of the following criteria:

  * Primary tumor and regional nodes resected with clear surgical margins and no evidence of extrahepatic disease
  * Unresected primary tumor with plans to resect the primary tumor before randomization
  * Unresected primary tumor with plans to resect the primary tumor and the liver metastases in a single surgical procedure performed after randomization
* No unresected primary tumor in the colon or rectum with significant symptoms related to obstruction or that will require radiotherapy

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy ≥ 5 years (excluding the diagnosis of metastatic CRC)
* absolute neutrophil count (ANC) ≥ 1,200/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Total bilirubin ≤ upper limit of normal (ULN)
* aspartate aminotransferase (AST) ≤ 5.0 times ULN
* Alkaline phosphatase ≤ 5.0 times ULN
* Serum creatinine ≤ ULN OR calculated creatinine clearance ≥ 30 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 180 days after completion of study treatment
* Considered a potential candidate for a major hepatic surgical procedure
* No grade 3 or 4 anorexia, grade 3 nausea, or vomiting ≥ grade 2 (per CTCAE v4.0) related to metastatic disease
* No paresthesias, peripheral sensory neuropathy, or peripheral motor neuropathy ≥ grade 2 per Common Toxicity Criteria for Adverse Effects (CTCAE) v4.0 (patients with grade 2 neuropathy who will receive FOLFIRI are eligible)
* No uncontrolled high BP defined as systolic BP ≥ 160 mm Hg OR diastolic BP ≥ 100 mm Hg, with or without antihypertensive medication (patients with initial BP elevations are eligible provided initiation or adjustment of BP medication lowers pressure to meet this criteria)
* Documented history of congestive heart failure requiring chronic medical therapy
* No active inflammatory bowel disease
* No active infection or chronic infection requiring chronic suppressive antibiotics
* No known bleeding diathesis or coagulopathy
* No symptomatic interstitial pneumonitis OR definitive evidence of interstitial pneumonitis described on CT scan, MRI, or chest x-ray in asymptomatic patients
* No other malignancies unless the patient is considered to be disease-free and has completed therapy for the malignancy ≥ 1 year ago

  * Patients with carcinoma in situ of the cervix, CRC in situ, melanoma in situ, or basal cell or squamous cell carcinoma of the skin diagnosed and treated at any time before study treatment are eligible
* No known Gilbert syndrome
* Not known to be homozygous for the UGT1A1 allele (for patients who will receive FOLFIRI chemotherapy)
* No prior serious hypersensitivity reaction to any of the agents administered as part of study treatment (determination of "serious" is at the investigator's discretion)
* No other serious concurrent medical condition that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to participate in the study, or cause a delay in the initiation of therapy (surgery or chemotherapy) longer than 4 weeks following randomization
* No psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements
* No pre-existing chronic hepatic disease (e.g., chronic active hepatitis, cirrhosis) that, in the opinion of the investigator and hepatic surgeon, would limit the patient's ability to undergo hepatic metastasectomy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No previous hepatic-directed therapy, including hepatic resection and/or ablation, hepatic arterial infusion therapy, or hepatic radiotherapy

  * Patients who have only had an incision or excisional biopsy are eligible
* No previous chemotherapy or any other systemic therapy for metastatic colorectal cancer (CRC)
* No prior or concurrent portal vein embolization or other hepatic preconditioning techniques
* At least 30 days since prior investigational products
* No intent to use ablation to treat any hepatic lesion
* No concurrent therapeutic doses of coumadin or equivalent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (283):
- United States (283):
  - Kaiser Permanente - Deer Valley, Antioch, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Kaiser Permanente - Moanalua Medical Center and Clinic, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Cancer Center - West Lakes, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - Ochsner Health Center - Covington, Covington, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Harry and Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton MD, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Berkshire Hematology Oncology, PC, Pittsfield, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls Medical Group, PA, Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Comprehensive Cancer Care, PC, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Nalitt Cancer Institute at Staten Island University Hospital, Staten Island, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Riddle Memorial Hospital Cancer Center, Media, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Associates in Hematology-Oncology, PC at Crozer Regional Cancer Center, Upland, Pennsylvania
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Self Regional Cancer Center at Self Regional Medical Center, Greenwood, South Carolina
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Overlake Cancer Center at Overlake Hospital Medical Center, Bellevue, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Postoperative Chemotherapy | Arm 2: Perioperative Chemotherapy
Started | 6 | 3
Completed | 0 | 0
Not Completed | 6 | 3
Not completed — Study terminated due to low accrual | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Postoperative Chemotherapy: Postoperative chemotherapy
- Perioperative Chemotherapy: Perioperative chemotherapy
- Total: Total of all reporting groups
Arm/Group | Postoperative Chemotherapy | Perioperative Chemotherapy | Total
Number analyzed (Participants) | 6 | 3 | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (14.9) | 55 (13.9) | 61 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival (RFS)
Description: Time to recurrence or death
Time Frame: From study entry until the date of recurrence or death or for a maximum of 5 years.
Arm/Group | Arm 1: Postoperative Chemotherapy | Arm 2: Perioperative Chemotherapy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: RFS of Patients Event-free
Time Frame: From study entry until the date of recurrence or for a maximum of 6 months.
Reporting Status: Not Posted

3. Secondary Outcome: Overall Survival
Time Frame: From study entry until the time of death or for a maximum of 5 years.
Reporting Status: Not Posted

4. Secondary Outcome: The Difference in R0 and Combined R0 + R1 Resection Rates Between the Two Arms.
Time Frame: Assessed at the time of surgery
Reporting Status: Not Posted

5. Secondary Outcome: Frequencies of Selected Postoperative Surgical Complications and Other Adverse Events Within 30 Days of Surgery
Time Frame: Assessed within 30 days from the time of surgery
Reporting Status: Not Posted

6. Secondary Outcome: Frequencies of Adverse Events as Assessed by the NCI CTCAE v4.0
Time Frame: From study entry through 3 months after the last treatment dose.
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Participants at Risk includes any patient who submitted an AE form.
Arm/Group | Postoperative Chemotherapy | Perioperative Chemotherapy
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/2
Other Adverse Events (participants affected / at risk) | 3/5 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Postoperative Chemotherapy (N=5) | Perioperative Chemotherapy (N=2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Postoperative Chemotherapy (N=5) | Perioperative Chemotherapy (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less